CLINICAL TRIAL: NCT02248753
Title: Acute Cardioversion Versus Wait And See-approach for Symptomatic Atrial Fibrillation in the Emergency Department (RACE 7 ACWAS-trial)
Brief Title: Acute Cardioversion Versus Wait And See-approach for Symptomatic Atrial Fibrillation in the Emergency Department
Acronym: RACE 7 ACWAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL47065.068.13; 837002524 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Electrical cardioversion; Pharmacological cardioversion; Rhythm control; Rate control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide; Electric Countershock; Metoprolol; Verapamil; Digoxin; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Active Comparator): Pharmacological cardioversion and/or electrical cardioversion
  Interventions: Drug: Pharmacological cardioversion - Flecainide; Procedure: Electrical cardioversion; Drug: Pharmacological cardioversion - Amiodarone
- Wait-and-see Approach (Experimental): Rate control drugs only (metoprolol, verapamil or digoxin)
  Interventions: Drug: Metoprolol; Drug: Verapamil; Drug: Digoxin

INTERVENTIONS:
Drug: Pharmacological cardioversion - Flecainide
  Other Names: Flecainide; Tambocor
  Arms: Standard Care
Procedure: Electrical cardioversion
  Arms: Standard Care
Drug: Metoprolol
  Other Names: Selokeen
  Arms: Wait-and-see Approach
Drug: Verapamil
  Other Names: Isoptin
  Arms: Wait-and-see Approach
Drug: Digoxin
  Other Names: Lanoxin
  Arms: Wait-and-see Approach
Drug: Pharmacological cardioversion - Amiodarone
  Other Names: Amiodarone; Cordarone
  Arms: Standard Care

SUMMARY:
A symptomatic episode of the heart rhythm disorder 'atrial fibrillation' (AF) is a frequent reason for visits to the emergency department. Currently, in the majority of cases, immediate (electrical or pharmacological) cardioversion is chosen, while atrial fibrillation terminates spontaneously in 70% of the cases within 24 hours. A wait-and-see approach with rate-control medication only, and when needed cardioversion within 48 hours of onset of symptoms, could be effective, safe and more cost-effective than current standard of care and could lead to a higher quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ECG with atrial fibrillation at the emergency department
* Heart rate > 70bpm
* Symptoms most probable due to atrial fibrillation
* Duration of symptoms < 36 hours
* > 18 years of age
* Able and willing to sign informed consent
* Able and willing to use MyDiagnostick

Exclusion Criteria:

* Signs of myocardial infarction on ECG
* Hemodynamic instability (systolic blood pressure < 100mm Hg, heart rate > 170 bpm)
* Presence of pre-excitation syndrome
* History of Sick Sinus Syndrome
* History of unexplained syncope
* History of persistent AF (episode of AF lasting more than 48 hours)
* Acute heart failure
* Currently enrolled in another clinical trial
* Deemed unsuitable for participation by attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
12-lead ECG | 4 weeks
  Presence of sinus rhythm on ECG

SECONDARY OUTCOMES:
Time to conversion to sinus rhythm (Holter monitor) | 48 hours
  Intervention group only
Quality of life (SF-36) | Baseline, 4 weeks, 6 months, 12 months
One-year follow-up of Major Adverse Cerebrovascular or Cardiovascular Events | One year
Time to first recurrence of Atrial Fibrillation | 1 month
  Monitoring through handheld device
Total health care and societal costs | 1 year
Quality of Life (AFEQT) | Baseline, 4 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Harry J Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (15):
- Netherlands (15):
  - VU University Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Zuyderland Medical Center, Heerlen
  - Alrijne Hospital, Leiderdorp
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Hospital, Nieuwegein
  - Franciscus Gasthuis, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - HagaZiekenhuis, The Hague
  - St. Elisabeth - TweeSteden Hospital, Tilburg
  - Diakonessenhuis, Utrecht
  - VieCuri Medical Center, Venlo

REFERENCES:
- [Background] Dudink E, Essers B, Holvoet W, Weijs B, Luermans J, Ramanna H, Liem A, van Opstal J, Dekker L, van Dijk V, Lenderink T, Kamp O, Kulker L, Rienstra M, Kietselaer B, Alings M, Widdershoven J, Meeder J, Prins M, van Gelder I, Crijns H. Acute cardioversion vs a wait-and-see approach for recent-onset symptomatic atrial fibrillation in the emergency department: Rationale and design of the randomized ACWAS trial. Am Heart J. 2017 Jan;183:49-53. doi: 10.1016/j.ahj.2016.09.009. Epub 2016 Oct 2. PMID 27979041
- [Derived] van der Velden RMJ, Pluymaekers NAHA, Dudink EAMP, Luermans JGLM, Meeder JG, Heesen WF, Lenderink T, Widdershoven JWMG, Bucx JJJ, Rienstra M, Kamp O, van Opstal JM, Kirchhof CJHJ, van Dijk VF, Swart HP, Alings M, Van Gelder IC, Crijns HJGM, Linz D. Mobile health adherence for the detection of recurrent recent-onset atrial fibrillation. Heart. 2022 Dec 13;109(1):26-33. doi: 10.1136/heartjnl-2022-321346. PMID 36322782
- [Derived] Pluymaekers NAHA, Dudink EAMP, Luermans JGLM, Meeder JG, Lenderink T, Widdershoven J, Bucx JJJ, Rienstra M, Kamp O, Van Opstal JM, Alings M, Oomen A, Kirchhof CJ, Van Dijk VF, Ramanna H, Liem A, Dekker LR, Essers BAB, Tijssen JGP, Van Gelder IC, Crijns HJGM; RACE 7 ACWAS Investigators. Early or Delayed Cardioversion in Recent-Onset Atrial Fibrillation. N Engl J Med. 2019 Apr 18;380(16):1499-1508. doi: 10.1056/NEJMoa1900353. Epub 2019 Mar 18. PMID 30883054